CLINICAL TRIAL: NCT00226954
Title: Zoledronic Acid With Intermittent Hormonal Therapy in Patients With Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Sandy Srinivas, PI, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROS0001; 78869; NCT00226954; PROS0001
Record Dates: First submitted 2005-09-13; First posted 2005-09-27 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Urologic Neoplasms
MeSH Terms: conditions — Urologic Neoplasms | interventions — Zoledronic Acid

ARMS (1):
- Zoledronic Acid with Intermittent Hormonal Therapy (Experimental)
  Interventions: Drug: zoledronic acid

INTERVENTIONS:
Drug: zoledronic acid

SUMMARY:
Primary:

To determine the duration of use of zoledronic acid in improving Bone mineral density in patients with prostate cancer who are on hormones intermittently.

Secondary Objectives:

To describe the safety and tolerability at this dose and schedule

ELIGIBILITY:
Inclusion Criteria:Patients: Who are 18 years of age and older Who have histologically documented adenocarcinoma of prostate Who are currently receiving LHRH agonists KPS greater than 80%Life expectancy greater than 6 months Provide written consent pursuant to regulatory requirements prior to initiation of study procedure Exclusion Criteria:Exclusion Criteria: Patients: Any patient requiring continuous LHRH Any patient who has had an orchiectomy Any patient with painful bone metastases Who have received chemotherapy for prostate cancer Who have a abnormal serum creatine >2.5 Receiving any investigational drug within the last 28 days Severe uncontrolled infection, diabetes, cardiac disease Patients with fragility fractures, hyperparathyroidism, Pagets renal osteodystrophy will be excluded History of non compliance to medical regimens or unwillingness to return for medical visits

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2003-03; Primary Completion 2007-11 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
To determine the duration of use of zoledronic acid in improving Bone mineral density in patients with prostate cancer who are on hormones intermittently.

SECONDARY OUTCOMES:
To describe the safety and tolerability at this dose and schedule

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sandy Srinivas, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States